CLINICAL TRIAL: NCT04520048
Title: Exploratory Study. Endothelial Function and Vascular-tropic Biomarkers: Predictive Indicators of the Progression of Hypertensive Disorders in Pregnancy to Pre-eclampsia?
Brief Title: Vascular Biomarkers Predictive of the Progression From Hypertensive Disorders in Pregnancy to Preeclampsia in Pregnant Women
Acronym: BIOVASC-PreHTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APHP200237; 2019-A03207-50 (Other: IDRCB)
Record Dates: First submitted 2020-07-17; First posted 2020-08-20 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Hypertension Disorders in Pregnancy; Gestational Hypertension; Pre-Eclampsia
Keywords: Hypertension disorders in pregnancy; Gestational hypertension; Pre-eclampsia; Urinary endothelial microparticules; Endothelial dysfunction; Angiogenic biomarkers; Soluble Fms-like- tyrosine kinase 1; Placental Growth Factor; Vascular Endothelial Growth Factor; Microcirculation
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Women with a hypertension disorder in pregnancy and/or preeclampsia (Experimental): Pregnant patients from the 20th week of amenorrhea with the initial diagnosis of a hypertension disorder in pregnancy and/or preeclampsia. Patients in a stable state undergoing follow-up consultation (day hospital and week hospitalization)
  Interventions: Other: Determination of the UEMP levels; Procedure: Aortic central pressure and the carotid-femoral pulse wave velocity; Other: Vascular biomarker assay; Procedure: Measurement of the uterine artery diameter

INTERVENTIONS:
Other: Determination of the UEMP levels — Quantification of UEMP by flow cytometry in urine (10 ml) collected at 26 ± 2 week and 34th ± 2 week of amenorrhea.
Procedure: Aortic central pressure and the carotid-femoral pulse wave velocity — Measurement of the aortic central arterial pressure (systolic and diastolic arterial pressure) by applanation tonometry, and the index of aortic increase by applanation tonometry, the carotid-femoral pulse wave velocity using the SphygmoCor® system (PWV Medical) and/or Popmetre.
Other: Vascular biomarker assay — Plasma angiogenic biomarker levels determination using an immunoassay, including circulating sFlt-1, circulating PIGF, sFlt-1 / PIGF ratio, circulating VEGF, circulating soluble endoglin (sEng), other biomarkers assessment, including anti-angiotensin II receptor (AT1), circulating copeptin, circulating interleukin 17 (IL-17), Urinary Neutrophil Gelatinase-Associated Lipocalin (NGAL), as well as CEMP and CEC quantification using flow cytometry.
Procedure: Measurement of the uterine artery diameter — This measurement is added to the routine examination of the uterine artery. Bi-dimensional ultrasound imaging with angio-Doppler allows the study of the artery as the blood flow velocity and vessel diameter. Uterine artery Doppler pulsatility index (UtA-PI), mean flow velocity and diameter measurement could be calculated with Doppler instrument with software could determine instantaneous true mean blood flow velocity. Measurement is made by placing the cursor from outer edge to outer edge of the artery adventitia, on a cross-section and taking the largest diameter

SUMMARY:
Hypertension during pregnancy remains a leading cause of maternal and fetal morbidity and mortality. The frequency (5 to 10% of pregnancies) and potential severity of these diseases, both for the mother and the child, are reasons for standardizing and optimizing medical practices.

The cause of hypertension during pregnancy is quite complex, as it depends on a number of factors. Among the hypertensive disorders in pregnancy (HDP), the pathophysiology of pre-eclampsia (one of the most studied in terms of severity) remains poorly understood. The evolution of international guidelines in recent years has made it possible to distinguish various HDP, but schematically we distinguish two main entities by the existence of proteinuria from and after the 20th week of amenorrhea and by maternal-fetal complications, more serious in pre-eclampsia than in gestational hypertension.

Acute placental vasculature and blood flow abnormalities were observed during gestational hypertension and preeclampsia, and maybe due to generalized vascular endothelial activation and vasospasm resulting in systemic hypertension and organ hypoperfusion. Endothelial dysfunction (ED) and abnormal expression of several specific blood biomarkers are now well accepted as characteristics of preeclampsia as a leader.

However, the progression of any HDP to preeclampsia is possible, but difficult to predict. By way of example, among between 15 and 40 % of gestational hypertension cases progress to preeclampsia, suggesting that it is the same worsening disease.

ED could be pre-existing (chronic, white-coat or masked hypertension) but also at the origin of gestational hypertension (unclassified hypertension, transient pregnancy hypertension), and subsequent development of preeclampsia through an imbalance between pro- and anti-angiogenic factors.

An imbalance of pro-angiogenic and anti-angiogenic proteins can testify to ED, as can adequate levels of endothelial microparticles.

The main objective of this research is to assess the presence of urinary endothelial microparticles in stable pregnant women with hypertensive disorder of pregnancy as a marker for the occurrence of pre-eclampsia during pregnancy.

DETAILED DESCRIPTION:
Hypertension in pregnancy is defined by PAS ≥140 mmHg and/or PAD ≥ 90 mmHg, mild to moderate hypertension by PAS = 140-159 mmHg and/or PAD = 90-109 mmHg and severe hypertension by PAS ≥ 160 mmHg and/or PAD ≥ 110 mmHg.

Definitions of hypertensive disorders in pregnancy have evolved considerably. We know that during gestational hypertension (GE) there is no pathologic elevation of proteinuria (after 20 weeks of amenorrhea). Preeclampsia (PE) is defined as high blood pressure (controlled or uncontrolled) associated with proteinuria discovered after the 20th week of amenorrhea.

The cause of hypertension and pathophysiology during pregnancy and in particular of preeclampsia remains poorly understood. Endothelial dysfunction and abnormal blood levels of several biomarkers are associated with PE, such as: soluble Fms-like- tyrosine kinase 1 (sFlt-1), Placental Growth Factor (PIGF) and Vascular Endothelial Growth Factor (VEGF). VEGF is of particular importance due to its direct vasodilating effect at systemic level through its interaction with nitric oxide (NO). There is a bi-directional regulation between VEGF and NO, which has direct implications for endothelium, capillary permeability and angiogenesis. sFlt-1 (circulating form of VEGF receptor) has the property of neutraliting the growth factors VEGF and PIGF. Inhibition of VEGF has a known biological effect on endothelial function in adults and is believed to be a key factor in explaining elevated blood pressure. This has been demonstrated in patients undergoing anti-angiogenic therapy in combination with chemotherapy. Other biomarkers of preeclampsia are less known and could be involved in pathophysiological mechanisms; mainly hypervolemia, renal dysfunction and activation of inflammation. The progression of gestational hypertension to preeclampsia is difficult to predict; between 15 and 40 % of gestational hypertension cases progress to preeclampsia, suggesting that it is a single worsening disease. Preeclampsia is known to be one of the few diseases in which acute placental abnormalities manifest at the mother's vascular and renal system levels. These abnormalities are attributable to generalized vascular endothelial activation and vasospasm, resulting in hypertension and hypoperfusion of organs.

Endothelial dysfunction could be at the origin of HDP as gestational hypertension, and subsequently itself contribute to the subsequent development of severe forms such preeclampsia through an imbalance between pro- and anti-angiogenic factors likely in relation with increased oxidative stress.

It is now accepted that angiogenic biomarkers (such as soluble fms-like tyrosine kinase 1, Placenta growth factor and soluble endoglin) contribute to endothelial dysfunction through VEGF antagonizing among others. The dosage of these angiogenic biomarkers in the maternal bloodstream is highly predictive and significantly abnormal from the 23th week of amenorrhea on average, and with a maximum peak between the 32th and 36th week of amenorrhea.

Endothelial microparticles (EMPs) are involved in intracellular communication and produced in normal pregnancy and in PE. The renal damage associated with PE and the potential role of extracellular vesicles are in the main adverse mechanisms that distinguish the different types of hypertension in pregnancy.

Adequate levels of circulating endothelial microparticles (CEMP), circulating endothelial cells (CECs), and endothelial progenitor cells most likely play an important role in the development and regulation of the vasculature during pregnancy, but the exact role in the pathogenesis of PE is unknown.

These endothelial microparticles (EMPs) reflects systemic endothelial damage and can also be measured in urine by flow cytometry. In general, in hypertensive patients, there is peritubular capillary loss (PCL) and it can be measured by these EMPs. Urinary (not blood) MP levels correlate directly with renal hypoxia and fibrosis and inversely with cortical perfusion. Therefore, the level of EMPs could be useful as "new biomarkers" of intrarenal capillary loss. However, only a few in-depth studies in the field of hypertension in pregnancy have focused on this issue.

The main objective is to assess whether the presence of urinary endothelial microparticles (UEMP) in the pregnant woman in a stable condition with discovery of HDP is a marker of the occurrence of preeclampsia later during pregnancy.

The investigators further explore a possible correlation of alteration of UEMP to other biomarkers of pre-eclampsia endothelial dysfunction and vascular involvement in pregnancy hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a hypertension disorder in pregnancy and/or preeclampsia from the 20th amenorrhea week until the 26th ± 2 amenorrhea week.
* Age between 18 and 40 years old.
* Having given written consent.
* Patients affiliated to a social security scheme.

Exclusion Criteria:

* Presence of pathologies interfering in a major way with vascular parameters: known multicomplicated diabetes treated before pregnancy, hypercholesterolemia known (or LDL>130 mg/dl), multicomplicated connectivitis, proven cardiovascular disease (ischemic heart disease, stroke, arteriopathy of the lower limbs, heart failure), pre-existing known renal failure (serum creatinine >125 µmol/L) and/or pre-existing proteinuria ≥ 300 mg/24h).
* Cardiac arrhythmia.
* Hepatitis C, HIV infection (assay performed within 6 months prior to diagnosis of pre-eclampsia).
* Recent history of venous (pulmonary embolism, phlebitis) or arterial (myocardial infarction, unstable angina, stroke, transient ischemic attack), thrombotic event ≤ 3 months.
* Patient already engaged in a therapeutic protocol.
* Patients under legal protective measures.
* Patients receiving State Medical Assistance.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 110 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in the UEMP levels between 26th ± 2 week and 34th ± 2 week of pregnancy. | change between the 26th ± 2 week of amenorrhea and 34th ± 2 week of amenorrhea
  Quantification of UEMP by flow cytometry in urine collected at 26 ± 2 week and 34th ± 2 week of amenorrhea.

SECONDARY OUTCOMES:
Change in circulating levels of soluble Fms-like tyrosine kinase (sFlt-1) between 26 weeks and 34 weeks of pregnancy | change between the 26th ± 2 week and 34th ± 2 week of amenorrhea
  Determining of circulating levels of sFlt-1 in the serum of patients using un immunoassay
Change in circulating Placental Growth factor (PIGF) between 26 weeks and 34 weeks of pregnancy | change between the 26th ± 2 week and 34th ± 2 week of amenorrhea
  Determining of circulating levels of PlGF in the serum of patients using un immunoassay
Change in circulating levels of vascular endothelial growth factors (VEGF) between 26 weeks and 34 weeks of pregnancy | change between the 26th ± 2 week and 34th ± 2 week of amenorrhea
  Determining of circulating levels of VEGF in the serum of patients using un immunoassay
Change in circulating levels of soluble endogline (sEng) between 26 weeks and 34 weeks of pregnancy | change between the 26th ± 2 week and 34th ± 2 week of amenorrhea
  Determining of circulating levels of sEng-1 in the serum of patients using un immunoassay
Change in angiotensin II receptor (AT1) between 26 weeks and 34 weeks of pregnancy | change between the 26th ± 2 week and 34th ± 2 week of amenorrhea
  Measurement of the angiotensin II receptor (AT1) levels in the serum of patients using un immunoassay
Change in the circulating Copetid levels between 26 weeks and 34 weeks of pregnancy | change between the 26th ± 2 week and 34th ± 2 week of amenorrhea
  Measurement of circulating Copetid levels in the serum of patients using un immunoassay
Change in circulating levels of Interleukin IL-17 between 26 weeks and 34 weeks of pregnancy | change between the 26th ± 2 week and 34th ± 2 week of amenorrhea
  Determining of circulating levels of Interleukin IL-17 in the serum of patients using un immunoassay
Change in urinary levels of Neutrophil Gelatinase-Associated Lipocalin (NGAL) between 26 weeks and 34 weeks of pregnancy | change between the 26th ± 2 week and 34th ± 2 week of amenorrhea
  Determining of urinary levels of NGAL using un immunoassay
Change in circulating Endothelial Microparticle Levels between 26 weeks and 34 weeks of pregnancy | change between the 26th ± 2 week and 34th ± 2 week of amenorrhea
  Determining of the blood levels of CEMP using flow cytometry
Change in circulating Endothelial Celle Levels between 26 weeks and 34 weeks of pregnancy | change between the 26th ± 2 week and 34th ± 2 week of amenorrhea
  Determining of the blood levels of CEC using flow cytometry
Change in central aortic blood pressure between 26 weeks and 34 weeks of pregnancy | change between the 26th ± 2 week and 34th ± 2 week of amenorrhea
  Measurement of the aortic central arterial pressure (systolic and diastolic arterial pressure) by applanation tonometry, and the index of aortic increase by applanation tonometry, using the SphygmoCor® system (PWV Medical) and/or Popmetre.
Change in carotid-femoral pulse wave velocity between 26 weeks and 34 weeks of pregnancy | change between the 26th ± 2 week and 34th ± 2 week of amenorrhea
  Measurement of the carotid-femoral pulse wave velocity using the SphygmoCor® system (PWV Medical)
Change in the uterine artery diameter between 26 weeks and 34 weeks of pregnancy | change between the 26th ± 2 week and 34th ± 2 week of amenorrhea
  Determining of the uterine artery diameter by bi-dimensional ultrasound imaging with angio-Doppler allows the study of the artery as the blood flow velocity and vessel diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Marilucy LOPEZ-SUBLET, MD, Principal Investigator — AP-HP Avicenne Hospital, Department of Internal Medicine, ESH Hypertension European Excellence Centre
Locations (3):
- France (3):
  - AP-HP Avicenne Hospital, Department of internal medicine, Bobigny, Seine Saint Denis
  - AP-HP Jean Verdier Hospital, Gynecology and Obstetrics Department, Bondy, Seine Saint Denis
  - AP-HP Laribosière Hospital, Gynecology and Obstetrics Department, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomopoulos C, Hitij JB, De Backer T, Gkaliagkousi E, Kreutz R, Lopez-Sublet M, Marketou M, Mihailidou AS, Olszanecka A, Pechere-Bertschi A, Perez MP, Persu A, Piani F, Socrates T, Stolarz-Skrzypek K, Cifkova R. Management of hypertensive disorders in pregnancy: a Position Statement of the European Society of Hypertension Working Group 'Hypertension in Women'. J Hypertens. 2024 Jul 1;42(7):1109-1132. doi: 10.1097/HJH.0000000000003739. Epub 2024 Apr 11. PMID 38690949
- [Background] Mancia G, Kreutz R, Brunstrom M, Burnier M, Grassi G, Januszewicz A, Muiesan ML, Tsioufis K, Agabiti-Rosei E, Algharably EAE, Azizi M, Benetos A, Borghi C, Hitij JB, Cifkova R, Coca A, Cornelissen V, Cruickshank JK, Cunha PG, Danser AHJ, Pinho RM, Delles C, Dominiczak AF, Dorobantu M, Doumas M, Fernandez-Alfonso MS, Halimi JM, Jarai Z, Jelakovic B, Jordan J, Kuznetsova T, Laurent S, Lovic D, Lurbe E, Mahfoud F, Manolis A, Miglinas M, Narkiewicz K, Niiranen T, Palatini P, Parati G, Pathak A, Persu A, Polonia J, Redon J, Sarafidis P, Schmieder R, Spronck B, Stabouli S, Stergiou G, Taddei S, Thomopoulos C, Tomaszewski M, Van de Borne P, Wanner C, Weber T, Williams B, Zhang ZY, Kjeldsen SE. 2023 ESH Guidelines for the management of arterial hypertension The Task Force for the management of arterial hypertension of the European Society of Hypertension: Endorsed by the International Society of Hypertension (ISH) and the European Renal Association (ERA). J Hypertens. 2023 Dec 1;41(12):1874-2071. doi: 10.1097/HJH.0000000000003480. Epub 2023 Sep 26. PMID 37345492
- [Background] Wu P, Haththotuwa R, Kwok CS, Babu A, Kotronias RA, Rushton C, Zaman A, Fryer AA, Kadam U, Chew-Graham CA, Mamas MA. Preeclampsia and Future Cardiovascular Health: A Systematic Review and Meta-Analysis. Circ Cardiovasc Qual Outcomes. 2017 Feb;10(2):e003497. doi: 10.1161/CIRCOUTCOMES.116.003497. Epub 2017 Feb 22. PMID 28228456
- [Background] SFHTA, M.-V.C.e.a., HTA et Grossesse. Consensus d'Experts de la Société Françaises d'Hypertension Artérielle. Consensus d'Experts avec le partenariat du Collège National des Gynécologues et Obstétriciens Français. 2015, Decembre: p. 1-5.
- [Background] Levine RJ, Maynard SE, Qian C, Lim KH, England LJ, Yu KF, Schisterman EF, Thadhani R, Sachs BP, Epstein FH, Sibai BM, Sukhatme VP, Karumanchi SA. Circulating angiogenic factors and the risk of preeclampsia. N Engl J Med. 2004 Feb 12;350(7):672-83. doi: 10.1056/NEJMoa031884. Epub 2004 Feb 5. PMID 14764923
- [Background] Noori M, Donald AE, Angelakopoulou A, Hingorani AD, Williams DJ. Prospective study of placental angiogenic factors and maternal vascular function before and after preeclampsia and gestational hypertension. Circulation. 2010 Aug 3;122(5):478-87. doi: 10.1161/CIRCULATIONAHA.109.895458. Epub 2010 Jul 19. PMID 20644016
- [Background] Kleinrouweler CE, Wiegerinck MM, Ris-Stalpers C, Bossuyt PM, van der Post JA, von Dadelszen P, Mol BW, Pajkrt E; EBM CONNECT Collaboration. Accuracy of circulating placental growth factor, vascular endothelial growth factor, soluble fms-like tyrosine kinase 1 and soluble endoglin in the prediction of pre-eclampsia: a systematic review and meta-analysis. BJOG. 2012 Jun;119(7):778-87. doi: 10.1111/j.1471-0528.2012.03311.x. Epub 2012 Mar 20. PMID 22433027
- [Background] Karumanchi SA. Angiogenic Factors in Preeclampsia: From Diagnosis to Therapy. Hypertension. 2016 Jun;67(6):1072-9. doi: 10.1161/HYPERTENSIONAHA.116.06421. Epub 2016 Apr 11. No abstract available. PMID 27067718
- [Background] Verlohren S, Perschel FH, Thilaganathan B, Droge LA, Henrich W, Busjahn A, Khalil A. Angiogenic Markers and Cardiovascular Indices in the Prediction of Hypertensive Disorders of Pregnancy. Hypertension. 2017 Jun;69(6):1192-1197. doi: 10.1161/HYPERTENSIONAHA.117.09256. Epub 2017 May 1. PMID 28461601
- [Background] Bouloumie A, Schini-Kerth VB, Busse R. Vascular endothelial growth factor up-regulates nitric oxide synthase expression in endothelial cells. Cardiovasc Res. 1999 Mar;41(3):773-80. doi: 10.1016/s0008-6363(98)00228-4. PMID 10435050
- [Background] Dulak J, Jozkowicz A, Dembinska-Kiec A, Guevara I, Zdzienicka A, Zmudzinska-Grochot D, Florek I, Wojtowicz A, Szuba A, Cooke JP. Nitric oxide induces the synthesis of vascular endothelial growth factor by rat vascular smooth muscle cells. Arterioscler Thromb Vasc Biol. 2000 Mar;20(3):659-66. doi: 10.1161/01.atv.20.3.659. PMID 10712388
- [Background] Yang JC, Haworth L, Sherry RM, Hwu P, Schwartzentruber DJ, Topalian SL, Steinberg SM, Chen HX, Rosenberg SA. A randomized trial of bevacizumab, an anti-vascular endothelial growth factor antibody, for metastatic renal cancer. N Engl J Med. 2003 Jul 31;349(5):427-34. doi: 10.1056/NEJMoa021491. PMID 12890841
- [Background] Mourad JJ, des Guetz G, Debbabi H, Levy BI. Blood pressure rise following angiogenesis inhibition by bevacizumab. A crucial role for microcirculation. Ann Oncol. 2008 May;19(5):927-34. doi: 10.1093/annonc/mdm550. Epub 2007 Dec 4. PMID 18056916
- [Background] Artunc-Ulkumen B, Guvenc Y, Goker A, Gozukara C. Relationship of neutrophil gelatinase-associated lipocalin (NGAL) and procalcitonin levels with the presence and severity of the preeclampsia. J Matern Fetal Neonatal Med. 2015 Nov;28(16):1895-900. doi: 10.3109/14767058.2014.972926. Epub 2014 Oct 29. PMID 25283849
- [Background] Yesil A, Kanawati A, Helvacioglu C, Kaya C, Ozgun CG, Cengiz H. Identification of patients at risk for preeclampsia with the use of uterine artery Doppler velocimetry and copeptin. J Matern Fetal Neonatal Med. 2017 Nov;30(22):2763-2768. doi: 10.1080/14767058.2016.1262841. Epub 2016 Dec 7. PMID 27868455
- [Background] Sun IO, Santelli A, Abumoawad A, Eirin A, Ferguson CM, Woollard JR, Lerman A, Textor SC, Puranik AS, Lerman LO. Loss of Renal Peritubular Capillaries in Hypertensive Patients Is Detectable by Urinary Endothelial Microparticle Levels. Hypertension. 2018 Nov;72(5):1180-1188. doi: 10.1161/HYPERTENSIONAHA.118.11766. PMID 30354805
- [Background] Szpera-Gozdziewicz A, Breborowicz GH. Endothelial dysfunction in the pathogenesis of pre-eclampsia. Front Biosci (Landmark Ed). 2014 Jan 1;19(5):734-46. doi: 10.2741/4240. PMID 24389217
- [Background] Hayman R, Brockelsby J, Kenny L, Baker P. Preeclampsia: the endothelium, circulating factor(s) and vascular endothelial growth factor. J Soc Gynecol Investig. 1999 Jan-Feb;6(1):3-10. PMID 10065419
- [Background] Pagani F, Cantaluppi V. Renal Injury During Preclampsia: Role of Extracellular Vesicles. Nephron. 2019;143(3):197-201. doi: 10.1159/000502456. Epub 2019 Aug 21. PMID 31434070
- [Background] Debbabi H, Bonnin P, Ducluzeau PH, Leftheriotis G, Levy BI. Noninvasive assessment of endothelial function in the skin microcirculation. Am J Hypertens. 2010 May;23(5):541-6. doi: 10.1038/ajh.2010.10. Epub 2010 Feb 18. PMID 20168305
- [Background] Chambers JC, Fusi L, Malik IS, Haskard DO, De Swiet M, Kooner JS. Association of maternal endothelial dysfunction with preeclampsia. JAMA. 2001 Mar 28;285(12):1607-12. doi: 10.1001/jama.285.12.1607. PMID 11268269
- [Background] Davis KR, Ponnampalam J, Hayman R, Baker PN, Arulkumaran S, Donnelly R. Microvascular vasodilator response to acetylcholine is increased in women with pre-eclampsia. BJOG. 2001 Jun;108(6):610-4. doi: 10.1111/j.1471-0528.2001.00144.x. PMID 11426896
- [Background] Ramsay JE, Stewart F, Greer IA, Sattar N. Microvascular dysfunction: a link between pre-eclampsia and maternal coronary heart disease. BJOG. 2003 Nov;110(11):1029-31. PMID 14592589
- [Background] Agatisa PK, Ness RB, Roberts JM, Costantino JP, Kuller LH, McLaughlin MK. Impairment of endothelial function in women with a history of preeclampsia: an indicator of cardiovascular risk. Am J Physiol Heart Circ Physiol. 2004 Apr;286(4):H1389-93. doi: 10.1152/ajpheart.00298.2003. PMID 15020302
- [Background] Khan F, Belch JJ, MacLeod M, Mires G. Changes in endothelial function precede the clinical disease in women in whom preeclampsia develops. Hypertension. 2005 Nov;46(5):1123-8. doi: 10.1161/01.HYP.0000186328.90667.95. Epub 2005 Oct 17. PMID 16230524
- [Background] Report of the National High Blood Pressure Education Program Working Group on High Blood Pressure in Pregnancy. Am J Obstet Gynecol. 2000 Jul;183(1):S1-S22. PMID 10920346
- [Background] Hauth JC, Ewell MG, Levine RJ, Esterlitz JR, Sibai B, Curet LB, Catalano PM, Morris CD. Pregnancy outcomes in healthy nulliparas who developed hypertension. Calcium for Preeclampsia Prevention Study Group. Obstet Gynecol. 2000 Jan;95(1):24-8. doi: 10.1016/s0029-7844(99)00462-7. PMID 10636496
- [Background] Hnat MD, Sibai BM, Caritis S, Hauth J, Lindheimer MD, MacPherson C, VanDorsten JP, Landon M, Miodovnik M, Paul R, Meis P, Thurnau G, Dombrowski M; National Institute of Child Health and Human Development Network of Maternal-Fetal Medicine-Units. Perinatal outcome in women with recurrent preeclampsia compared with women who develop preeclampsia as nulliparas. Am J Obstet Gynecol. 2002 Mar;186(3):422-6. doi: 10.1067/mob.2002.120280. PMID 11904601
- [Background] Cain MA, Salemi JL, Tanner JP, Kirby RS, Salihu HM, Louis JM. Pregnancy as a window to future health: maternal placental syndromes and short-term cardiovascular outcomes. Am J Obstet Gynecol. 2016 Oct;215(4):484.e1-484.e14. doi: 10.1016/j.ajog.2016.05.047. Epub 2016 Jun 2. PMID 27263996
- [Background] Buchbinder A, Sibai BM, Caritis S, Macpherson C, Hauth J, Lindheimer MD, Klebanoff M, Vandorsten P, Landon M, Paul R, Miodovnik M, Meis P, Thurnau G; National Institute of Child Health and Human Development Network of Maternal-Fetal Medicine Units. Adverse perinatal outcomes are significantly higher in severe gestational hypertension than in mild preeclampsia. Am J Obstet Gynecol. 2002 Jan;186(1):66-71. doi: 10.1067/mob.2002.120080. PMID 11810087
- [Background] Myatt L, Roberts JM. Preeclampsia: Syndrome or Disease? Curr Hypertens Rep. 2015 Nov;17(11):83. doi: 10.1007/s11906-015-0595-4. PMID 26362531
- [Background] Hod T, Cerdeira AS, Karumanchi SA. Molecular Mechanisms of Preeclampsia. Cold Spring Harb Perspect Med. 2015 Aug 20;5(10):a023473. doi: 10.1101/cshperspect.a023473. PMID 26292986
- [Background] Powe CE, Levine RJ, Karumanchi SA. Preeclampsia, a disease of the maternal endothelium: the role of antiangiogenic factors and implications for later cardiovascular disease. Circulation. 2011 Jun 21;123(24):2856-69. doi: 10.1161/CIRCULATIONAHA.109.853127. No abstract available. PMID 21690502
- [Background] Hirashima C, Ohkuchi A, Takahashi K, Suzuki H, Yoshida M, Ohmaru T, Eguchi K, Ariga H, Matsubara S, Suzuki M. Gestational hypertension as a subclinical preeclampsia in view of serum levels of angiogenesis-related factors. Hypertens Res. 2011 Feb;34(2):212-7. doi: 10.1038/hr.2010.212. Epub 2010 Nov 4. PMID 21048778
- [Background] Allen RE, Rogozinska E, Cleverly K, Aquilina J, Thangaratinam S. Abnormal blood biomarkers in early pregnancy are associated with preeclampsia: a meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2014 Nov;182:194-201. doi: 10.1016/j.ejogrb.2014.09.027. Epub 2014 Sep 22. PMID 25305662
- [Background] Lam C, Lim KH, Karumanchi SA. Circulating angiogenic factors in the pathogenesis and prediction of preeclampsia. Hypertension. 2005 Nov;46(5):1077-85. doi: 10.1161/01.HYP.0000187899.34379.b0. Epub 2005 Oct 17. PMID 16230516
- [Background] Motta-Mejia C, Kandzija N, Zhang W, Mhlomi V, Cerdeira AS, Burdujan A, Tannetta D, Dragovic R, Sargent IL, Redman CW, Kishore U, Vatish M. Placental Vesicles Carry Active Endothelial Nitric Oxide Synthase and Their Activity is Reduced in Preeclampsia. Hypertension. 2017 Aug;70(2):372-381. doi: 10.1161/HYPERTENSIONAHA.117.09321. Epub 2017 Jun 12. PMID 28607124
- [Background] Rana S, Powe CE, Salahuddin S, Verlohren S, Perschel FH, Levine RJ, Lim KH, Wenger JB, Thadhani R, Karumanchi SA. Angiogenic factors and the risk of adverse outcomes in women with suspected preeclampsia. Circulation. 2012 Feb 21;125(7):911-9. doi: 10.1161/CIRCULATIONAHA.111.054361. Epub 2012 Jan 18. PMID 22261192
- [Background] Lely AT, Salahuddin S, Holwerda KM, Karumanchi SA, Rana S. Circulating lymphangiogenic factors in preeclampsia. Hypertens Pregnancy. 2013;32(1):42-9. doi: 10.3109/10641955.2012.697953. Epub 2012 Sep 7. PMID 22957504
- [Background] Turpin CA, Sakyi SA, Owiredu WK, Ephraim RK, Anto EO. Association between adverse pregnancy outcome and imbalance in angiogenic regulators and oxidative stress biomarkers in gestational hypertension and preeclampsia. BMC Pregnancy Childbirth. 2015 Aug 25;15:189. doi: 10.1186/s12884-015-0624-y. PMID 26303772
- [Background] Mannaerts D, Faes E, Goovaerts I, Stoop T, Cornette J, Gyselaers W, Spaanderman M, Van Craenenbroeck EM, Jacquemyn Y. Flow-mediated dilation and peripheral arterial tonometry are disturbed in preeclampsia and reflect different aspects of endothelial function. Am J Physiol Regul Integr Comp Physiol. 2017 Nov 1;313(5):R518-R525. doi: 10.1152/ajpregu.00514.2016. Epub 2017 Aug 9. PMID 28794106
- [Background] Matsubara K, Abe E, Matsubara Y, Kameda K, Ito M. Circulating endothelial progenitor cells during normal pregnancy and pre-eclampsia. Am J Reprod Immunol. 2006 Aug;56(2):79-85. doi: 10.1111/j.1600-0897.2006.00387.x. PMID 16836609
- [Background] Redman CW, Sargent IL. Microparticles and immunomodulation in pregnancy and pre-eclampsia. J Reprod Immunol. 2007 Dec;76(1-2):61-7. doi: 10.1016/j.jri.2007.03.008. Epub 2007 May 4. PMID 17482271
- [Background] Guller S, Tang Z, Ma YY, Di Santo S, Sager R, Schneider H. Protein composition of microparticles shed from human placenta during placental perfusion: Potential role in angiogenesis and fibrinolysis in preeclampsia. Placenta. 2011 Jan;32(1):63-9. doi: 10.1016/j.placenta.2010.10.011. Epub 2010 Nov 11. PMID 21074265
- [Background] VanWijk MJ, Nieuwland R, Boer K, van der Post JA, VanBavel E, Sturk A. Microparticle subpopulations are increased in preeclampsia: possible involvement in vascular dysfunction? Am J Obstet Gynecol. 2002 Aug;187(2):450-6. doi: 10.1067/mob.2002.124279. PMID 12193942
- [Background] van der Post JA, Lok CA, Boer K, Sturk A, Sargent IL, Nieuwland R. The functions of microparticles in pre-eclampsia. Semin Thromb Hemost. 2011 Mar;37(2):146-52. doi: 10.1055/s-0030-1270342. Epub 2011 Mar 2. PMID 21370216
- [Background] Gonzalez-Quintero VH, Jimenez JJ, Jy W, Mauro LM, Hortman L, O'Sullivan MJ, Ahn Y. Elevated plasma endothelial microparticles in preeclampsia. Am J Obstet Gynecol. 2003 Aug;189(2):589-93. doi: 10.1067/s0002-9378(03)00469-1. PMID 14520240
- [Background] Prochazka M, Prochazkova J, Lubusky M, Pilka R, Ulehlova J, Michalec I, Polak P, Kacerovsky M, Slavik L. Markers of endothelial activation in preeclampsia. Clin Lab. 2015;61(1-2):39-46. PMID 25807636
- [Background] Ling L, Huang H, Zhu L, Mao T, Shen Q, Zhang H. Evaluation of plasma endothelial microparticles in pre-eclampsia. J Int Med Res. 2014 Feb;42(1):42-51. doi: 10.1177/0300060513504362. Epub 2013 Dec 6. PMID 24319051
- [Background] Petrozella L, Mahendroo M, Timmons B, Roberts S, McIntire D, Alexander JM. Endothelial microparticles and the antiangiogenic state in preeclampsia and the postpartum period. Am J Obstet Gynecol. 2012 Aug;207(2):140.e20-6. doi: 10.1016/j.ajog.2012.06.011. Epub 2012 Jun 11. PMID 22840727
- [Background] Salem M, Kamal S, El Sherbiny W, Abdel Aal AA. Flow cytometric assessment of endothelial and platelet microparticles in preeclampsia and their relation to disease severity and Doppler parameters. Hematology. 2015 Apr;20(3):154-9. doi: 10.1179/1607845414Y.0000000178. Epub 2014 Jul 7. PMID 25001068
- [Background] Alijotas-Reig J, Palacio-Garcia C, Farran-Codina I, Ruiz-Romance M, Llurba E, Vilardell-Tarres M. Circulating cell-derived microparticles in severe preeclampsia and in fetal growth restriction. Am J Reprod Immunol. 2012 Feb;67(2):140-51. doi: 10.1111/j.1600-0897.2011.01072.x. Epub 2011 Oct 13. PMID 21992597
- [Background] Anim-Nyame N, Ghosh A, Freestone N, Arrigoni FI. Relationship between insulin resistance and circulating endothelial cells in pre-eclampsia. Gynecol Endocrinol. 2015 Oct;31(10):788-91. doi: 10.3109/09513590.2015.1065477. Epub 2015 Jul 14. PMID 26172933
- [Background] Wallukat G, Homuth V, Fischer T, Lindschau C, Horstkamp B, Jupner A, Baur E, Nissen E, Vetter K, Neichel D, Dudenhausen JW, Haller H, Luft FC. Patients with preeclampsia develop agonistic autoantibodies against the angiotensin AT1 receptor. J Clin Invest. 1999 Apr;103(7):945-52. doi: 10.1172/JCI4106. PMID 10194466
- [Background] Signore C, Mills JL, Qian C, Yu K, Lam C, Epstein FH, Karumanchi SA, Levine RJ. Circulating angiogenic factors and placental abruption. Obstet Gynecol. 2006 Aug;108(2):338-44. doi: 10.1097/01.AOG.0000216014.72503.09. PMID 16880304
- [Background] Zhou CC, Irani RA, Zhang Y, Blackwell SC, Mi T, Wen J, Shelat H, Geng YJ, Ramin SM, Kellems RE, Xia Y. Angiotensin receptor agonistic autoantibody-mediated tumor necrosis factor-alpha induction contributes to increased soluble endoglin production in preeclampsia. Circulation. 2010 Jan 26;121(3):436-44. doi: 10.1161/CIRCULATIONAHA.109.902890. Epub 2010 Jan 11. PMID 20065159
- [Background] Antonios TF, Nama V, Wang D, Manyonda IT. Microvascular remodelling in preeclampsia: quantifying capillary rarefaction accurately and independently predicts preeclampsia. Am J Hypertens. 2013 Sep;26(9):1162-9. doi: 10.1093/ajh/hpt087. Epub 2013 Jun 11. PMID 23757401
- [Background] Wu J, Thabet SR, Kirabo A, Trott DW, Saleh MA, Xiao L, Madhur MS, Chen W, Harrison DG. Inflammation and mechanical stretch promote aortic stiffening in hypertension through activation of p38 mitogen-activated protein kinase. Circ Res. 2014 Feb 14;114(4):616-25. doi: 10.1161/CIRCRESAHA.114.302157. Epub 2013 Dec 17. PMID 24347665
- [Background] Madhur MS, Lob HE, McCann LA, Iwakura Y, Blinder Y, Guzik TJ, Harrison DG. Interleukin 17 promotes angiotensin II-induced hypertension and vascular dysfunction. Hypertension. 2010 Feb;55(2):500-7. doi: 10.1161/HYPERTENSIONAHA.109.145094. Epub 2009 Dec 28. PMID 20038749
- [Background] Darmochwal-Kolarz D, Michalak M, Kolarz B, Przegalinska-Kalamucka M, Bojarska-Junak A, Sliwa D, Oleszczuk J. The Role of Interleukin-17, Interleukin-23, and Transforming Growth Factor-beta in Pregnancy Complicated by Placental Insufficiency. Biomed Res Int. 2017;2017:6904325. doi: 10.1155/2017/6904325. Epub 2017 Jun 15. PMID 28698875
- [Background] Borgel D, Chocron R, Grimaud M, Philippe A, Chareyre J, Brakta C, Lasne D, Bonnet D, Toubiana J, Angoulvant F, Desvages M, Renolleau S, Smadja DM, Oualha M. Endothelial Dysfunction as a Component of Severe Acute Respiratory Syndrome Coronavirus 2-Related Multisystem Inflammatory Syndrome in Children With Shock. Crit Care Med. 2021 Nov 1;49(11):e1151-e1156. doi: 10.1097/CCM.0000000000005093. PMID 34049308
- [Background] Smadja DM, Mentzer SJ, Fontenay M, Laffan MA, Ackermann M, Helms J, Jonigk D, Chocron R, Pier GB, Gendron N, Pons S, Diehl JL, Margadant C, Guerin C, Huijbers EJM, Philippe A, Chapuis N, Nowak-Sliwinska P, Karagiannidis C, Sanchez O, Kumpers P, Skurnik D, Randi AM, Griffioen AW. COVID-19 is a systemic vascular hemopathy: insight for mechanistic and clinical aspects. Angiogenesis. 2021 Nov;24(4):755-788. doi: 10.1007/s10456-021-09805-6. Epub 2021 Jun 28. PMID 34184164
- [Background] Papageorghiou AT, Yu CK, Erasmus IE, Cuckle HS, Nicolaides KH. Assessment of risk for the development of pre-eclampsia by maternal characteristics and uterine artery Doppler. BJOG. 2005 Jun;112(6):703-9. doi: 10.1111/j.1471-0528.2005.00519.x. PMID 15924523
- [Background] Ray JG, Vermeulen MJ, Schull MJ, Redelmeier DA. Cardiovascular health after maternal placental syndromes (CHAMPS): population-based retrospective cohort study. Lancet. 2005 Nov 19;366(9499):1797-803. doi: 10.1016/S0140-6736(05)67726-4. PMID 16298217
- [Background] Rich-Edwards JW. The predictive pregnancy: what complicated pregnancies tell us about mother's future cardiovascular risk. Circulation. 2012 Mar 20;125(11):1336-8. doi: 10.1161/CIRCULATIONAHA.112.093872. Epub 2012 Feb 21. No abstract available. PMID 22354939
- [Background] Brown MA, Buddle ML. What's in a name? Problems with the classification of hypertension in pregnancy. J Hypertens. 1997 Oct;15(10):1049-54. doi: 10.1097/00004872-199715100-00001. No abstract available. PMID 9350577
- [Background] Saudan P, Brown MA, Buddle ML, Jones M. Does gestational hypertension become pre-eclampsia? Br J Obstet Gynaecol. 1998 Nov;105(11):1177-84. doi: 10.1111/j.1471-0528.1998.tb09971.x. PMID 9853766
- [Background] Davis GK, Mackenzie C, Brown MA, Homer CS, Holt J, McHugh L, Mangos G. Predicting transformation from gestational hypertension to preeclampsia in clinical practice: a possible role for 24 hour ambulatory blood pressure monitoring. Hypertens Pregnancy. 2007;26(1):77-87. doi: 10.1080/10641950601147952. PMID 17454220
- [Background] Palomaki GE, Haddow JE, Haddow HR, Salahuddin S, Geahchan C, Cerdeira AS, Verlohren S, Perschel FH, Horowitz G, Thadhani R, Karumanchi SA, Rana S. Modeling risk for severe adverse outcomes using angiogenic factor measurements in women with suspected preterm preeclampsia. Prenat Diagn. 2015 Apr;35(4):386-93. doi: 10.1002/pd.4554. Epub 2015 Feb 4. PMID 25641027
- [Background] Moore Simas TA, Crawford SL, Solitro MJ, Frost SC, Meyer BA, Maynard SE. Angiogenic factors for the prediction of preeclampsia in high-risk women. Am J Obstet Gynecol. 2007 Sep;197(3):244.e1-8. doi: 10.1016/j.ajog.2007.06.030. PMID 17826405
- [Background] Maynard SE, Crawford SL, Bathgate S, Yan J, Robidoux L, Moore M, Moore Simas TA. Gestational angiogenic biomarker patterns in high risk preeclampsia groups. Am J Obstet Gynecol. 2013 Jul;209(1):53.e1-9. doi: 10.1016/j.ajog.2013.03.017. Epub 2013 Mar 18. PMID 23517919